CLINICAL TRIAL: NCT01169818
Title: Asian Treat to Target Lantus Study: A Randomized, Multicentre, Multinational, Open-Label, Parallel-Group, 24-Week Phase IV Study Evaluating the Effectiveness and Safety of Physician Versus Patient-led Initiation and Titration of Insulin Glargine in Type 2 Diabetes Mellitus
Brief Title: Evaluation of the Effectiveness and Safety of Physician Versus Patient-led of Insulin Glargine Initiation and Titration in Type 2 Diabetes Mellitus
Acronym: ATLAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LANTU_R_04889; U1111-1116-2247 (Other: UTN)
Record Dates: First submitted 2010-07-22; First posted 2010-07-26 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

ARMS (2):
- Intervention group (Experimental): Initiation on a fixed dose of insulin glargine, then subjects will self-adjusted their basal insulin dose every 3 days
  Interventions: Drug: Insulin Glargine
- Usual standard of care group (Active Comparator): Initiation on a fixed dose of insulin glargine, then basal insulin dose is adjusted at each visit by a physician
  Interventions: Drug: Insulin Glargine

INTERVENTIONS:
Drug: Insulin Glargine — Pharmaceutical form: solution for injection
  Route of administration: subcutaneous
  Dose regimen: initial: once a day in the evening at bedtime. Titration will occur each time the middle FPG (Fasting Plasma Glucose) value is above target
  Other Names: Solostar

SUMMARY:
Primary Objective:

To compare patient-led titration (intervention group) versus physician-led titration (usual standard of care) in optimizing the clinical use of insulin glargine in an Asian population of patients with Type 2 diabetes mellitus (T2DM) uncontrolled on oral antidiabetic drugs (OADs).

Secondary Objectives:

To determine the difference in glycemic control, safety, quality of life and treatment satisfaction between patient-led titration and usual care.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosed with T2DM duration of T2DM > 2 years
2. Insulin naïve
3. Continuous treatment with stable doses of 2 OADs (sulphonylureas, biguanides, alpha-glucosidase inhibitors, DPP-IV inhibitors, and glinides) for > three months prior to randomization
4. HbA1c levels 7% and 11 %
5. Body mass index (BMI) 20 and 40 kg/m2
6. Willing and able to perform blood glucose monitoring using a blood glucose meter

Exclusion criteria:

1. Diabetes other than type 2 diabetes (e.g. secondary to pancreatic disorders, drug or chemical agent intake),
2. Current or previous use of insulin (except for previous treatment of gestational diabetes or brief treatment with insulin for < 1 week),
3. Current treatment with thiazolidinediones,
4. Current or previous use (within the last 3 months) of GLP-1 receptor agonists or GLP-1 analogues,
5. Current or previous (within the last 3 months) use of any treatment for weight lost,
6. Active proliferative diabetic retinopathy,
7. Patient without any history of eye examination in the past 6 months,
8. Treatment with systemic corticosteroids in the 3 months prior to study entry,
9. Currently receiving treatment with monoamine oxidase inhibitors,
10. Currently receiving treatment with non-selective -blockers,
11. Treatment with any investigational product and/or device in the 2 months prior to study entry,
12. Likelihood of requiring treatment during the study period with drugs not permitted by the clinical trial protocol,
13. History of ketoacidosis or hyperosmolar hyperglycemic state,
14. History of stroke, myocardial infarction, angina pectoris, coronary artery bypass graft or percutaneous transluminal coronary angioplasty within the previous 12 months,
15. History of congestive heart failure,
16. History of hypoglycemia unawareness,
17. Unexplained hypoglycemia in the past 6 months,
18. Impaired renal function defined as, but not limited to, serum creatinine 1.5 mg/dL (133 mol/L) males or 1.4 mg/dL (124 mol/L) females or presence of macroproteinuria (>2gr/day),
19. Active liver disease (alanine transaminase ALAT greater than two times the upper limit of the reference range, as defined by the local laboratory),
20. Have any condition (including known substance or alcohol abuse or psychiatric disorder) that precludes the patient from following and completing the study protocol,
21. Had a blood transfusion or severe blood loss within the 3 months before screening, or have known hemoglobinopathy, hemolytic anemia or sickle cell anemia,
22. Known hypersensitivity / intolerance to insulin glargine or any of its excipients,
23. History of pancreatitis,
24. Currently undergoing therapy or planned radiological examinations requiring the administration of contrasting agents for malignancy (other than non-metastatic / early stage basal cell or squamous cell carcinoma),
25. Pregnant or lactating women (women of childbearing potential must have a negative pregnancy test at study entry and a medically approved contraception method),
26. Any medical condition that may have an influence on HbA1c rate.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 555 (Actual)
Dates: Start 2010-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change (decrease) in mean hemoglobin glycosylated (HbA1c) level | from week 0 (baseline) to week 24 (end of study)

SECONDARY OUTCOMES:
Percentage of patients achieving HbA1c levels < 7.0% without experiencing severe hypoglycemia | from week 0 (baseline) to week 24 (end of study)
Percentage of patients achieving target HbA1c levels (< 7.0% and <6.5%) | from week 0 (baseline) to week 24 (end of study)
Number of patients having a drop of 1% in HbA1c levels and/or a drop of at least 0.5%. | from week 0 (baseline) to week 24 (end of study)
Mean change in Fasting Plasma glucose (FPG) and Post Prandial blood Glucose (PPG) | from week 0 (baseline) to week 24 (end of study)
Evolution of Blood Glucose profiles | from week 0 (baseline) to week 24 (end of study)
Incidence of symptomatic hypoglycemia | from week 0 (baseline) to week 24 (end of study)
Incidence of nocturnal hypoglycemia | from week 0 (baseline) to week 24 (end of study)
Incidence of asymptomatic hypoglycemia | from week 0 (baseline) to week 24 (end of study)
Mean change in body weight in patients | from week 0 (baseline) to week 24 (end of study)
Mean insulin dose | from week 0 (baseline) to week 24 (end of study)
PROMs (patient reported outcome measures) scores from the DTSQs/c (diabetes treatment satisfaction questionnaire status) and EQ-5D (European quality of life - 5 dimensions) | from week 0 (baseline) to week 24 (end of study)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (6):
- Administrative office, Shanghai, China
- Administrative office, Mumbai, India
- Administrative office, Tokyo, Japan
- Administrative office, Karachi, Pakistan
- Administrative office, Makati City, Philippines
- Administrative office, Moscow, Russia

REFERENCES:
- [Background] ATLAS Study Group. Titration of Insulin Glargine in Patients with Type 2 Diabetes Mellitus in Asia: Physician- Versus Patient-Led? Rationale of the Asian Treat to Target Lantus Study (ATLAS). Diabetes Technol Ther. 2011 Jan;13(1):67-72. doi: 10.1089/dia.2010.0170. PMID 21175274
- [Derived] Garg SK, Admane K, Freemantle N, Odawara M, Pan CY, Misra A, Jarek-Martynowa IR, Abbas-Raza S, Mirasol RC, Perfetti R. Patient-led versus physician-led titration of insulin glargine in patients with uncontrolled type 2 diabetes: a randomized multinational ATLAS study. Endocr Pract. 2015 Feb;21(2):143-57. doi: 10.4158/EP14079.OR. PMID 25297660